CLINICAL TRIAL: NCT00996801
Title: A Phase IIb, Randomized, Double-Blind, Placebo- and Active-Controlled, Dose-Range-Finding Study to Evaluate the Effects of MK-5442 on Bone Mineral Density (BMD) in the Treatment of Osteoporosis in Postmenopausal Women Previously Treated With an Oral Bisphosphonate
Brief Title: MK-5442 in the Treatment of Osteoporosis in Postmenopausal Women Previously Treated With an Oral Bisphosphonate (MK-5442-012)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5442-012; 2009-014729-18 (EudraCT Number); CTRI/2010/091/000258 (Registry Identifier: CTRI)
Record Dates: First submitted 2009-10-15; First posted 2009-10-16 (Estimated); Results first posted 2012-11-16 (Estimated); Last update posted 2016-01-22 (Estimated); Status verified 2016-01

CONDITIONS: Osteoporosis; Postmenopausal Osteoporosis
MeSH Terms: conditions — Osteoporosis; Osteoporosis, Postmenopausal | interventions — JTT 305; Alendronate; Cholecalciferol; Calcium Carbonate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Placebo (Placebo Comparator): Participants received either matching placebo to alendronate (administered orally, once-weekly) or matching placebo to MK-5442 (administered orally, once-daily) for 12 months. Participants also received supplemental vitamin D3 and calcium (as needed) during treatment.
  Interventions: Drug: Placebo to MK-5442; Drug: Vitamin D3; Drug: Calcium carbonate; Drug: Placebo to Alendronate
- MK-5442 5 mg (Experimental): Participants received 5 mg of MK-5442 (orally, once-daily) plus matching placebo to alendronate (administered orally, once-weekly) for 12 months. Participants also received supplemental vitamin D3 and calcium (as needed) during treatment.
  Interventions: Drug: MK-5442; Drug: Vitamin D3; Drug: Calcium carbonate; Drug: Placebo to Alendronate
- MK-5442 7.5 mg (Experimental): Participants received 7.5 mg of MK-5442 (orally, once-daily) plus matching placebo to alendronate (administered orally, once-weekly) for 12 months. Participants also received supplemental vitamin D3 and calcium (as needed) during treatment.
  Interventions: Drug: MK-5442; Drug: Vitamin D3; Drug: Calcium carbonate; Drug: Placebo to Alendronate
- MK-5442 10 mg (Experimental): Participants received 10 mg of MK-5442 (orally, once-daily) plus matching placebo to alendronate (administered orally, once-weekly) for 12 months. Participants also received supplemental vitamin D3 and calcium (as needed) during treatment.
  Interventions: Drug: MK-5442; Drug: Vitamin D3; Drug: Calcium carbonate; Drug: Placebo to Alendronate
- MK-5442 15 mg (Experimental): Participants received 15 mg of MK-5442 (orally, once-daily) plus matching placebo to alendronate (administered orally, once-weekly) for 12 months. Participants also received supplemental vitamin D3 and calcium (as needed) during treatment.
  Interventions: Drug: MK-5442; Drug: Vitamin D3; Drug: Calcium carbonate; Drug: Placebo to Alendronate
- Alendronate 70 mg (Active Comparator): Participants received 70 mg alendronate (orally, once-weekly) plus matching placebo to MK-5442 (administered orally, once-daily) for 12 months. Participants also received supplemental vitamin D3 and calcium (as needed) during treatment.
  Interventions: Drug: Placebo to MK-5442; Drug: Alendronate Sodium; Drug: Vitamin D3; Drug: Calcium carbonate

INTERVENTIONS:
Drug: MK-5442 — MK-5442 tablets (randomized to a dose of 5, 7.5, 10 or 15 mg) taken orally, once-daily, for 12 months
  Arms: MK-5442 10 mg; MK-5442 15 mg; MK-5442 5 mg; MK-5442 7.5 mg
Drug: Placebo to MK-5442 — Matching placebo to MK-5442 taken orally, once-daily, for 12 months
  Arms: Alendronate 70 mg; Placebo
Drug: Alendronate Sodium — Alendronate tablets 70 mg, taken orally, once-weekly, for 12 months
  Other Names: FOSAMAX®
  Arms: Alendronate 70 mg
Drug: Vitamin D3 — Vitamin D3 (cholecalciferol) administered orally, at a dose of 5600 IU (two tablets, 2800 IU each), once-weekly for 12 months
  Other Names: Cholecalciferol
Drug: Calcium carbonate — Participants who qualify (those who have a calcium intake of less than 1200 mg/day) will receive oral supplemental calcium carbonate, at a dose of either 400 mg or 500 mg, once-daily, for 12 months
Drug: Placebo to Alendronate — Placebo to alendronate once-weekly for 12 months
  Arms: MK-5442 10 mg; MK-5442 15 mg; MK-5442 5 mg; MK-5442 7.5 mg; Placebo

SUMMARY:
This study seeks to demonstrate that additional gain in bone mineral density (BMD) can be achieved by switching to MK-5442 from an oral bisphosphonate in participants who have been receiving oral bisphosphonate therapy for at least 3 years.

DETAILED DESCRIPTION:
The study was originally planned for a duration of 2 years and included efficacy analysis of a 15 mg MK-5442 treatment arm. Amendment 1 of the protocol eliminated the 2nd year of the study as well the 15-mg arm. Enrollment into the 15-mg MK-5442 arm was stopped as a result of the amendment and all participants who had been randomly assigned to the MK-5442 15-mg treatment arm were discontinued from the study.

ELIGIBILITY:
Inclusion Criteria:

* Taking oral bisphosphonate treatment for osteoporosis for at least 3 of the past 4 years. At present, and for the past 12 months, treated with alendronate
* Bone Mineral Density (BMD) T-score that is ≤ -1.5 at one or more of the following anatomic sites; lumbar spine, femoral neck, trochanter, and total hip, AND a BMD T-score at all of these sites that is ≥ -4.0, AND a history of at least one fragility fracture, OR, a BMD T-score that is ≤ -2.5 at one or more of the following anatomic sites; lumbar spine, femoral neck, trochanter, and total hip, AND a BMD T-score at all of these sites that is ≥ -4.0
* Postmenopausal for at least 5 years

Exclusion Criteria:

* Obesity (ie, weight greater than 250 pounds) that prohibits the use of dual-emission X-ray absorptiometry (DXA)
* Received intravenous (IV) bisphosphonates, fluoride treatment at a dose >1 mg/day for more than 2 weeks, strontium, growth hormone, a cathepsin K (CTSK) inhibitor, or a receptor activator of nuclear factor kappa-B ligand (RANKL) inhibitor at any time in the past
* Use of oral bisphosphonates other than alendronate in the last 12 months, parathyroid hormone (PTH) in the last 24 months, cyclosporin for more than 2 weeks in the last 6 months, heparin in the last 2 weeks, or anabolic steroids or glucocorticoids for more than 2 weeks in the past 6 months
* Use of estrogen with or without progestin or a selective estrogen receptor modulator (SERM) in the last 6 months or calcitonin in the last 30 days
* Has used pioglitazone hydrochloride or rosiglitazone hydrochloride in the last 6 months
* Taking more than 10,000 International Units (IU) vitamin A daily or more than 5,000 IU vitamin D daily
* Has had a total thyroidectomy
* History of Paget's disease
* Has human immunodeficiency virus (HIV)
* History of cancer in the last 5 years, except certain skin or cervical cancers
* History of major upper gastrointestinal (GI) mucosal erosive disease
* Unable to adhere to dosing instructions for alendronate in regard to fasting and positioning
* Not ambulatory

Ages: 45 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 526 (Actual)
Dates: Start 2009-11; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

REFERENCES:
- [Result] Cosman F, Gilchrist N, McClung M, Foldes J, de Villiers T, Santora A, Leung A, Samanta S, Heyden N, McGinnis JP 2nd, Rosenberg E, Denker AE. A phase 2 study of MK-5442, a calcium-sensing receptor antagonist, in postmenopausal women with osteoporosis after long-term use of oral bisphosphonates. Osteoporos Int. 2016 Jan;27(1):377-86. doi: 10.1007/s00198-015-3392-7. Epub 2015 Nov 10. PMID 26556736
- [Derived] Saag K, Cosman F, De Villiers T, Langdahl B, Scott BB, Denker AE, Pong A, Santora AC. Early changes in bone turnover and bone mineral density after discontinuation of long-term oral bisphosphonates: a post hoc analysis. Osteoporos Int. 2021 Sep;32(9):1879-1888. doi: 10.1007/s00198-020-05785-3. Epub 2021 Feb 19. PMID 33606045

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | MK-5442 5 mg | MK-5442 7.5 mg | MK-5442 10 mg | MK-5442 15 mg | Alendronate 70 mg
Started | 88 | 88 | 88 | 87 | 88 (15-mg arm was discontinued as a result of Protocol Amendment 1.) | 87
Completed | 68 | 72 | 65 | 56 | 0 | 68
Not Completed | 20 | 16 | 23 | 31 | 88 | 19
Not completed — Adverse Event | 6 | 4 | 12 | 17 | 31 | 3
Not completed — Lack of Efficacy | 3 | 0 | 1 | 3 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 3 | 3 | 2
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Progressive Disease | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 3 | 4 | 1 | 2 | 3 | 4
Not completed — Study Terminated by Sponsor | 0 | 1 | 0 | 0 | 46 | 0
Not completed — Withdrawal by Subject | 8 | 6 | 9 | 5 | 5 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | MK-5442 5 mg | MK-5442 7.5 mg | MK-5442 10 mg | MK-5442 15 mg | Alendronate 70 mg | Total
Number analyzed (Participants) | 88 | 88 | 88 | 87 | 88 | 87 | 526
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.8 (7.8) | 66.5 (8.8) | 67.3 (7.1) | 68.2 (6.9) | 68.1 (7.4) | 66.9 (7.5) | 67.5 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88 | 88 | 88 | 87 | 88 | 87 | 526
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Least Squares Mean Percent Change From Baseline To Month 12 in Lumbar Spine Areal Bone Mineral Density (BMD)
Description: Areal bone mineral density (BMD) was measured using dual-energy X-ray absorptiometry (DXA) scanning technology. Scanning is performed with two X-ray beams with different energy levels which are aimed at the participant's bones. When soft tissue absorption is subtracted out, the BMD is determined from the absorption of each beam by bone.
  BMD = BMC / W, where BMD = bone mineral density in g/cm^2, BMC = bone mineral content in g/cm, and W = width at the scanned line in cm
Time Frame: Baseline and Month 12
Population: Full Analysis Set (FAS): participants who received at least one dose of study treatment, had at least one post-randomization observation, and who had baseline data.
  The MK-5442 15-mg treatment arm was discontinued as a result of Amendment 1 and thus no outcome analyses were performed.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Groups:
- Placebo: Participants received oral matching placebo for MK-5442 or alendronate, based on their randomization to active drug or comparator arm.
- MK-5442 5 mg: Participants were randomized to receive oral, once-daily MK-5442 5 mg and once-weekly matching placebo to alendronate for 12 months.
- MK-5442 7.5mg: Participants were randomized to receive oral, once-daily MK-5442 7.5 mg and once-weekly matching placebo to alendronate for 12 months.
- MK-5442 10 mg: Participants were randomized to receive oral, once-daily MK-5442 10 mg and once-weekly matching placebo to alendronate for 12 months.
- Alendronate 70 mg: Participants were randomized to receive oral, once-weekly alendronate 70 mg plus once-daily matching placebo to MK-5442 for 12 months.
Arm/Group | Placebo | MK-5442 5 mg | MK-5442 7.5mg | MK-5442 10 mg | Alendronate 70 mg
Number analyzed (Participants) | 81 | 82 | 79 | 78 | 79
percent change | -0.36 [-1.37 to 0.66] | -0.67 [-1.67 to 0.33] | -0.52 [-1.56 to 0.52] | -0.53 [-1.61 to 0.56] | 1.29 [0.25 to 2.33]
Statistical Analysis 1: Comparison: MK-5442 5 mg vs Alendronate 70 mg; Test type: Superiority or Other; p = 0.012, Longitudinal Data Analysis Model — The Type-I error rate over the multiple treatment dose comparisons were controlled by step-down Dunnett's test at the primary time point of Month 12, at an alpha level of 0.05, two-sided; Difference in Least Squares Means = -1.96, 95% CI 2-sided [-3.58 to -0.35]
Statistical Analysis 2: Comparison: MK-5442 7.5mg vs Alendronate 70 mg; Test type: Superiority or Other; p = 0.019, Longitudinal Data Analysis Model — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = -1.81, 95% CI 2-sided [-3.37 to -0.25]
Statistical Analysis 3: Comparison: MK-5442 10 mg vs Alendronate 70 mg; Test type: Superiority or Other; p = 0.019, Longitudinal Data Analysis Model — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = -1.82, 95% CI 2-sided [-3.23 to -0.41]

2. Secondary Outcome: Least Squares Mean Percent Change From Baseline to Month 12 in Total Hip Areal BMD
Description: Areal bone mineral density (BMD) was measured using DXA scanning technology. Scanning is performed with two X-ray beams with different energy levels which are aimed at the participant's bones. When soft tissue absorption is subtracted out, the BMD is determined from the absorption of each beam by bone.
  BMD = BMC / W, where BMD = bone mineral density in g/cm^2, BMC = bone mineral content in g/cm, and W = width at the scanned line in cm
Time Frame: Baseline and Month 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Groups:
- MK-5442 7.5 mg: Participants were randomized to receive oral, once-daily MK-5442 7.5 mg and once-weekly matching placebo to alendronate for 12 months.
Arm/Group | Placebo | MK-5442 5 mg | MK-5442 7.5 mg | MK-5442 10 mg | Alendronate 70 mg
Number analyzed (Participants) | 81 | 82 | 79 | 78 | 79
percent change | -1.44 [-2.24 to -0.65] | -2.18 [-2.97 to -1.39] | -2.16 [-2.98 to -1.33] | -1.66 [-2.52 to -0.80] | 0.46 [-0.36 to 1.29]
Statistical Analysis 1: Comparison: MK-5442 5 mg vs Alendronate 70 mg; Test type: Superiority or Other; p < 0.001, Longitudinal Data Analysis Model — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = -2.64, 95% CI 2-sided [-3.90 to -1.38]
Statistical Analysis 2: Comparison: MK-5442 7.5 mg vs Alendronate 70 mg; Test type: Superiority or Other; p < 0.001, Longitudinal Data Analysis Model — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = -2.62, 95% CI 2-sided [-3.83 to -1.40]
Statistical Analysis 3: Comparison: MK-5442 10 mg vs Alendronate 70 mg; Test type: Superiority or Other; p < 0.001, Longitudinal Data Analysis Model — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = -2.12, 95% CI 2-sided [-3.22 to -1.02]
Statistical Analysis 4: Comparison: Placebo vs MK-5442 5 mg; Test type: Superiority or Other; p = 0.376, Longitudinal Data Analysis Model — [p-value comment as in outcome 1, analysis 1]; Difference in Least Square Means = -0.74, 95% CI 2-sided [-1.99 to 0.52]
Statistical Analysis 5: Comparison: Placebo vs MK-5442 7.5 mg; Test type: Superiority or Other; p = 0.376, Longitudinal Data Analysis Model — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = -0.71, 95% CI 2-sided [-1.93 to 0.50]
Statistical Analysis 6: Comparison: Placebo vs MK-5442 10 mg; Test type: Superiority or Other; p = 0.699, Longitudinal Data Analysis Model — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = -0.22, 95% CI 2-sided [-1.32 to 0.88]

3. Secondary Outcome: Least Squares Mean Percent Change From Baseline to Month 12 in Femoral Neck Areal BMD
Description: as for outcome 2
Time Frame: Baseline and Month 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo | MK-5442 5 mg | MK-5442 7.5 mg | MK-5442 10 mg | Alendronate 70 mg
Number analyzed (Participants) | 81 | 82 | 79 | 78 | 79
percent change | -1.26 [-2.15 to -0.36] | -2.12 [-3.00 to -1.23] | -1.37 [-2.29 to -0.44] | -1.84 [-2.80 to -0.88] | -0.08 [-1.01 to 0.85]
Statistical Analysis 1: Comparison: MK-5442 5 mg vs Alendronate 70 mg; Test type: Superiority or Other; p = 0.002, Longitudinal Data Analysis Model — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = -2.04, 95% CI 2-sided [-3.43 to -0.64]
Statistical Analysis 2: Comparison: MK-5442 7.5 mg vs Alendronate 70 mg; Test type: Superiority or Other; p = 0.035, Longitudinal Data Analysis Model — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = -1.29, 95% CI 2-sided [-2.48 to -0.09]
Statistical Analysis 3: Comparison: MK-5442 10 mg vs Alendronate 70 mg; Test type: Superiority or Other; p = 0.009, Longitudinal Data Analysis Model — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = -1.76, 95% CI 2-sided [-3.14 to -0.38]
Statistical Analysis 4: Comparison: Placebo vs MK-5442 5 mg; Test type: Superiority or Other; p = 0.335, Longitudinal Data Analysis Model — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = -0.86, 95% CI 2-sided [-2.26 to 0.54]
Statistical Analysis 5: Comparison: Placebo vs MK-5442 7.5 mg; Test type: Superiority or Other; p = 0.857, Longitudinal Data Analysis Model — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = -0.11, 95% CI 2-sided [-1.30 to 1.08]
Statistical Analysis 6: Comparison: Placebo vs MK-5442 10 mg; Test type: Superiority or Other; p = 0.542, Longitudinal Data Analysis Model — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = -0.59, 95% CI 2-sided [-1.96 to 0.79]

4. Secondary Outcome: Least Squares Mean Percent Change From Baseline to Month 12 in Trochanter Areal BMD
Description: as for outcome 2
Time Frame: Baseline and Month 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo | MK-5442 5 mg | MK-5442 7.5 mg | MK-5442 10 mg | Alendronate 70 mg
Number analyzed (Participants) | 81 | 82 | 79 | 78 | 79
percent change | -0.30 [-1.35 to 0.76] | -1.56 [-2.60 to -0.52] | -1.50 [-2.59 to -0.41] | -1.52 [-2.66 to -0.38] | 1.68 [0.59 to 2.76]
Statistical Analysis 1: Comparison: MK-5442 5 mg vs Alendronate 70 mg; Test type: Superiority or Other; p < 0.001, Longitudinal Data Analysis Model — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = -3.24, 95% CI 2-sided [-4.91 to -1.57]
Statistical Analysis 2: Comparison: MK-5442 7.5 mg vs Alendronate 70 mg; Test type: Superiority or Other; p < 0.001, Longitudinal Data Analysis Model — [p-value comment as in outcome 1, analysis 1]; Difference in Least Square Means = -3.18, 95% CI 2-sided [-4.78 to -1.57]
Statistical Analysis 3: Comparison: MK-5442 10 mg vs Alendronate 70 mg; Test type: Superiority or Other; p < 0.001, Longitudinal Data Analysis Model — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = -3.20, 95% CI 2-sided [-4.66 to -1.74]
Statistical Analysis 4: Comparison: Placebo vs MK-5442 5 mg; Test type: Superiority or Other; p = 0.180, Longitudinal Data Analysis Model — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = -1.27, 95% CI 2-sided [-2.93 to 0.40]
Statistical Analysis 5: Comparison: Placebo vs MK-5442 7.5 mg; Test type: Superiority or Other; p = 0.180, Longitudinal Data Analysis Model — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = -1.20, 95% CI 2-sided [-2.81 to 0.40]
Statistical Analysis 6: Comparison: Placebo vs MK-5442 10 mg; Test type: Superiority or Other; p = 0.180, Longitudinal Data Analysis Model — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = -1.22, 95% CI 2-sided [-2.68 to 0.23]

5. Secondary Outcome: Least Squares Mean Percent Change From Baseline to Month 12 in Total Body Areal BMD
Description: as for outcome 2
Time Frame: Baseline and Month 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo | MK-5442 5 mg | MK-5442 7.5 mg | MK-5442 10 mg | Alendronate 70 mg
Number analyzed (Participants) | 68 | 75 | 70 | 74 | 72
percent change | -0.17 [-0.83 to 0.49] | -0.54 [-1.18 to 0.10] | -0.69 [-1.37 to -0.01] | -1.10 [-1.77 to -0.44] | 0.82 [0.15 to 1.48]
Statistical Analysis 1: Comparison: MK-5442 5 mg vs Alendronate 70 mg; Test type: Superiority or Other; p = 0.001, Longitudinal Data Analysis Model — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = -1.36, 95% CI 2-sided [-2.18 to -0.54]
Statistical Analysis 2: Comparison: MK-5442 7.5 mg vs Alendronate 70 mg; Test type: Superiority or Other; p = 0.001, Longitudinal Data Analysis Model — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = -1.51, 95% CI 2-sided [-2.46 to -0.55]
Statistical Analysis 3: Comparison: MK-5442 10 mg vs Alendronate 70 mg; Test type: Superiority or Other; p < 0.001, Longitudinal Data Analysis Model — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = -1.92, 95% CI 2-sided [-2.93 to -0.91]
Statistical Analysis 4: Comparison: Placebo vs MK-5442 5 mg; Test type: Superiority or Other; p = 0.383, Longitudinal Data Analysis Model — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = -0.37, 95% CI 2-sided [-1.21 to 0.46]
Statistical Analysis 5: Comparison: Placebo vs MK-5442 7.5 mg; Test type: Superiority or Other; p = 0.383, Longitudinal Data Analysis Model — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = -0.52, 95% CI 2-sided [-1.49 to 0.45]
Statistical Analysis 6: Comparison: Placebo vs MK-5442 10 mg; Test type: Superiority or Other; p = 0.084, Longitudinal Data Analysis Model — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = -0.94, 95% CI 2-sided [-1.96 to 0.09]

6. Secondary Outcome: Least Squares Mean Percent Change From Baseline to Month 12 in 1/3 Distal Forearm Areal BMD
Description: as for outcome 2
Time Frame: Baseline and Month 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo | MK-5442 5 mg | MK-5442 7.5 mg | MK-5442 10 mg | Alendronate 70 mg
Number analyzed (Participants) | 67 | 72 | 65 | 66 | 69
percent change | -0.54 [-1.54 to 0.46] | -1.38 [-2.36 to -0.40] | -0.92 [-1.95 to 0.12] | -2.01 [-3.05 to -0.98] | -0.91 [-1.92 to 0.10]
Statistical Analysis 1: Comparison: MK-5442 5 mg vs Alendronate 70 mg; Test type: Superiority or Other; p = 0.680, Longitudinal Data Analysis Model — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = -0.47, 95% CI 2-sided [-1.88 to 0.94]
Statistical Analysis 2: Comparison: MK-5442 7.5 mg vs Alendronate 70 mg; Test type: Superiority or Other; p = 0.993, Longitudinal Data Analysis Model — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = -0.01, 95% CI 2-sided [-1.30 to 1.28]
Statistical Analysis 3: Comparison: MK-5442 10 mg vs Alendronate 70 mg; Test type: Superiority or Other; p = 0.230, Longitudinal Data Analysis Model — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = -1.10, 95% CI 2-sided [-2.67 to 0.46]
Statistical Analysis 4: Comparison: Placebo vs MK-5442 5 mg; Test type: Superiority or Other; p = 0.333, Longitudinal Data Analysis Model — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = -0.84, 95% CI 2-sided [-2.29 to 0.61]
Statistical Analysis 5: Comparison: Placebo vs MK-5442 7.5 mg; Test type: Superiority or Other; p = 0.577, Longitudinal Data Analysis Model — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = -0.37, 95% CI 2-sided [-1.69 to 0.94]
Statistical Analysis 6: Comparison: Placebo vs MK-5442 10 mg; Test type: Superiority or Other; p = 0.078, Longitudinal Data Analysis Model — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = -1.47, 95% CI 2-sided [-3.07 to 0.12]

7. Secondary Outcome: Least Squares Mean Percent Change From Baseline to Month 12 in Trabecular Volumetric BMD (vBMD) of the Lumbar Spine
Description: vBMD was measured using quantitative computed tomography (QCT) in order to assess bone strength. Quantitative computed tomography is a three-dimensional non-projectional technique that quantifies trabecular and cortical BMD in the lumbar spine and hip as a true volumetric mineral density in g/cm^3.
Time Frame: Baseline and Month 12
Population: Full Analysis Set (FAS), QCT Subset: QCT was performed on a subset of the FAS (participants who received at least one dose of study treatment, had at least one post-randomization observation, and who had baseline data).
  The MK-5442 15-mg treatment arm was discontinued as a result of Amendment 1 and thus no outcome analyses were performed.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo | MK-5442 5 mg | MK-5442 7.5 mg | MK-5442 10 mg | Alendronate 70 mg
Number analyzed (Participants) | 45 | 58 | 49 | 49 | 43
percent change | 0.18 [-1.22 to 1.57] | -0.25 [-1.55 to 1.05] | 0.08 [-1.29 to 1.44] | 0.16 [-1.28 to 1.61] | 1.74 [0.21 to 3.26]
Statistical Analysis 1: Comparison: MK-5442 5 mg vs Alendronate 70 mg; Test type: Superiority or Other; p = 0.094, Longitudinal Data Analysis Model — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = -1.99, 95% CI 2-sided [-4.22 to 0.25]
Statistical Analysis 2: Comparison: MK-5442 7.5 mg vs Alendronate 70 mg; Test type: Superiority or Other; p = 0.157, Longitudinal Data Analysis Model — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = -1.66, 95% CI 2-sided [-3.82 to 0.50]
Statistical Analysis 3: Comparison: MK-5442 10 mg vs Alendronate 70 mg; Test type: Superiority or Other; p = 0.157, Longitudinal Data Analysis Model — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = -1.57, 95% CI 2-sided [-3.53 to 0.38]
Statistical Analysis 4: Comparison: Placebo vs MK-5442 5 mg; Test type: Superiority or Other; p = 0.937, Longitudinal Data Analysis Model — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = -0.43, 95% CI 2-sided [-2.61 to 1.76]
Statistical Analysis 5: Comparison: Placebo vs MK-5442 7.5 mg; Test type: Superiority or Other; p = 0.992, Longitudinal Data Analysis Model — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = -0.10, 95% CI 2-sided [-2.21 to 2.01]
Statistical Analysis 6: Comparison: Placebo vs MK-5442 10 mg; Test type: Superiority or Other; p = 0.992, Longitudinal Data Analysis Model — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = -0.01, 95% CI 2-sided [-1.93 to 1.90]

8. Secondary Outcome: Least Squares Mean Percent Change From Baseline to Month 12 in Trabecular Volumetric BMD of the Hip
Description: vBMD was measured using QCT in order to assess bone strength. QCT is a three-dimensional non-projectional technique that quantifies trabecular and cortical BMD in the lumbar spine and hip as a true volumetric mineral density in g/cm^3.
Time Frame: Baseline and Month 12
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo | MK-5442 5 mg | MK-5442 7.5 mg | MK-5442 10 mg | Alendronate 70 mg
Number analyzed (Participants) | 46 | 57 | 48 | 48 | 45
percent change | -0.02 [-1.41 to 1.36] | 0.76 [-0.53 to 2.05] | 0.81 [-0.57 to 2.18] | 0.27 [-1.16 to 1.71] | 1.23 [-0.23 to 2.70]
Statistical Analysis 1: Comparison: MK-5442 5 mg vs Alendronate 70 mg; Test type: Superiority or Other; p = 0.824, Longitudinal Data Analysis Model — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = -0.47, 95% CI 2-sided [-2.50 to 1.56]
Statistical Analysis 2: Comparison: MK-5442 7.5 mg vs Alendronate 70 mg; Test type: Superiority or Other; p = 0.824, Longitudinal Data Analysis Model — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = -0.42, 95% CI 2-sided [-2.28 to 1.43]
Statistical Analysis 3: Comparison: MK-5442 10 mg vs Alendronate 70 mg; Test type: Superiority or Other; p = 0.624, Longitudinal Data Analysis Model — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = -0.96, 95% CI 2-sided [-3.23 to 1.31]
Statistical Analysis 4: Comparison: Placebo vs MK-5442 5 mg; Test type: Superiority or Other; p = 0.700, Longitudinal Data Analysis Model — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = 0.78, 95% CI 2-sided [-1.25 to 2.82]
Statistical Analysis 5: Comparison: Placebo vs MK-5442 7.5 mg; Test type: Superiority or Other; p = 0.700, Longitudinal Data Analysis Model — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = 0.83, 95% CI 2-sided [-1.39 to 3.06]
Statistical Analysis 6: Comparison: Placebo vs MK-5442 10 mg; Test type: Superiority or Other; p = 0.759, Longitudinal Data Analysis Model — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = 0.30, 95% CI 2-sided [-1.60 to 2.19]

9. Secondary Outcome: Least Squares Mean Percent Change From Baseline to Month 12 in Cortical Volumetric BMD of the Lumbar Spine
Description: as for outcome 8
Time Frame: Baseline and Month 12
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo | MK-5442 5 mg | MK-5442 7.5 mg | MK-5442 10 mg | Alendronate 70 mg
Number analyzed (Participants) | 45 | 58 | 49 | 49 | 43
percent change | -0.67 [-15.01 to 13.66] | -3.41 [-16.35 to 9.52] | 14.66 [0.91 to 28.41] | -0.34 [-14.49 to 13.82] | 12.80 [-2.31 to 27.92]
Statistical Analysis 1: Comparison: MK-5442 5 mg vs Alendronate 70 mg; Test type: Superiority or Other; p = 0.227, Longitudinal Data Analysis Model — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = -16.22, 95% CI 2-sided [-39.15 to 6.72]
Statistical Analysis 2: Comparison: MK-5442 7.5 mg vs Alendronate 70 mg; Test type: Superiority or Other; p = 0.853, Longitudinal Data Analysis Model — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = 1.85, 95% CI 2-sided [-17.90 to 21.61]
Statistical Analysis 3: Comparison: MK-5442 10 mg vs Alendronate 70 mg; Test type: Superiority or Other; p = 0.327, Longitudinal Data Analysis Model — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = -13.14, 95% CI 2-sided [-35.67 to 9.39]
Statistical Analysis 4: Comparison: Placebo vs MK-5442 5 mg; Test type: Superiority or Other; p = 0.940, Longitudinal Data Analysis Model — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = -2.74, 95% CI 2-sided [-23.91 to 18.43]
Statistical Analysis 5: Comparison: Placebo vs MK-5442 7.5 mg; Test type: Superiority or Other; p = 0.273, Longitudinal Data Analysis Model — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = 15.33, 95% CI 2-sided [-7.86 to 38.52]
Statistical Analysis 6: Comparison: Placebo vs MK-5442 10 mg; Test type: Superiority or Other; p = 0.973, Longitudinal Data Analysis Model — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = 0.33, 95% CI 2-sided [-19.23 to 19.90]

10. Secondary Outcome: Least Squares Mean Percent Change From Baseline to Month 12 in Cortical Volumetric BMD of the Hip
Description: as for outcome 8
Time Frame: Baseline and Month 12
Population: Full Analysis Set (FAS), QCT Subset: QCT was performed on a subset of the FAS (participants who received at least one dose of study treatment, had at least one post-randomization observation, and who had baseline data).
  The MK-5442 15-mg treatment arm was discontinued as a result of Amendment 1 and thus no outcomes analyses were performed.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo | MK-5442 5 mg | MK-5442 7.5 mg | MK-5442 10 mg | Alendronate 70 mg
Number analyzed (Participants) | 46 | 57 | 48 | 48 | 45
percent change | 0.10 [-0.67 to 0.86] | -0.49 [-1.19 to 0.22] | -0.15 [-0.90 to 0.60] | -0.16 [-0.94 to 0.62] | 0.99 [0.19 to 1.78]
Statistical Analysis 1: Comparison: MK-5442 5 mg vs Alendronate 70 mg; Test type: Superiority or Other; p = 0.010, Longitudinal Data Analysis Model — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = -1.48, 95% CI 2-sided [-2.66 to -0.29]
Statistical Analysis 2: Comparison: MK-5442 7.5 mg vs Alendronate 70 mg; Test type: Superiority or Other; p = 0.053, Longitudinal Data Analysis Model — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = -1.14, 95% CI 2-sided [-2.29 to 0.01]
Statistical Analysis 3: Comparison: MK-5442 10 mg vs Alendronate 70 mg; Test type: Superiority or Other; p = 0.053, Longitudinal Data Analysis Model — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = -1.15, 95% CI 2-sided [-2.19 to -0.11]
Statistical Analysis 4: Comparison: Placebo vs MK-5442 5 mg; Test type: Superiority or Other; p = 0.509, Longitudinal Data Analysis Model — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = -0.58, 95% CI 2-sided [-1.77 to 0.60]
Statistical Analysis 5: Comparison: Placebo vs MK-5442 7.5 mg; Test type: Superiority or Other; p = 0.843, Longitudinal Data Analysis Model — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = -0.25, 95% CI 2-sided [-1.27 to 0.77]
Statistical Analysis 6: Comparison: Placebo vs MK-5442 10 mg; Test type: Superiority or Other; p = 0.843, Longitudinal Data Analysis Model — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = -0.26, 95% CI 2-sided [-1.43 to 0.92]

11. Secondary Outcome: Least Squares Mean Percent Change From Baseline to Month 12 in Urinary-N Telopeptides of Type 1 Collagen (u-NTx)
Description: Urinary, type I collagen, crosslinked N-telopeptide (uNTx) is a biomarker used to measure the rate of bone turnover found in urine.
  uNTx was expressed in units of nanomoles (nM) per bone collagen equivalents (BCE) per millimoles of creatinine (Cr) or nM/BCE/mM Cr
Time Frame: Baseline and Month 12
Population: Per Protocol Population: defined as the subset of the APaT population that excluded participants based on critical protocol violations.
  The MK-5442 15-mg treatment arm was discontinued as a result of Amendment 1 and thus no outcome analyses were performed.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo | MK-5442 5 mg | MK-5442 7.5 mg | MK-5442 10 mg | Alendronate 70 mg
Number analyzed (Participants) | 68 | 71 | 68 | 73 | 67
percent change | 63.64 [47.71 to 81.29] | 86.51 [68.86 to 106.01] | 83.32 [64.49 to 102.08] | 107.44 [86.65 to 130.54] | 0.18 [-9.45 to 10.83]
Statistical Analysis 1: Comparison: MK-5442 5 mg vs Alendronate 70 mg; Test type: Superiority or Other; p < 0.001, Constrained Longitudinal Data Analysis — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = 86.33, 95% CI 2-sided [64.87 to 108.29]
Statistical Analysis 2: Comparison: MK-5442 7.5 mg vs Alendronate 70 mg; Test type: Superiority or Other; p < 0.001, Constrained Longitudinal Data Analysis — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = 82.14, 95% CI 2-sided [63.00 to 101.66]
Statistical Analysis 3: Comparison: MK-5442 10 mg vs Alendronate 70 mg; Test type: Superiority or Other; p < 0.001, Constrained Longitudinal Data Analysis — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = 107.26, 95% CI 2-sided [82.03 to 133.23]
Statistical Analysis 4: Comparison: Placebo vs MK-5442 5 mg; Test type: Superiority or Other; p = 0.104, Constrained Longitudinal Data Analysis — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = 22.87, 95% CI 2-sided [-3.80 to 49.68]
Statistical Analysis 5: Comparison: Placebo vs MK-5442 7.5 mg; Test type: Superiority or Other; p = 0.123, Constrained Longitudinal Data Analysis — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = 18.68, 95% CI 2-sided [-5.11 to 42.56]
Statistical Analysis 6: Comparison: Placebo vs MK-5442 10 mg; Test type: Superiority or Other; p = 0.003, Constrained Longitudinal Data Analysis — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = 43.80, 95% CI 2-sided [12.85 to 75.06]

12. Secondary Outcome: Least Squares Mean Percent Change From Baseline to Month 12 in Serum C-Terminal Propeptide of Type 1 Collagen (s-CTx)
Description: C-Terminal Telopeptide Collagen I is used as a serum-marker of bone resorption in the assessment of osteoporosis and in measured in units of nanograms (n)/milliliter (ml).
Time Frame: Baseline and Month 12
Population: as for outcome 11
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo | MK-5442 5 mg | MK-5442 7.5 mg | MK-5442 10 mg | Alendronate 70 mg
Number analyzed (Participants) | 70 | 73 | 69 | 72 | 71
percent change | 165.80 [131.23 to 205.54] | 214.09 [173.92 to 260.15] | 227.07 [184.11 to 276.53] | 251.08 [204.31 to 305.04] | 26.78 [10.58 to 45.36]
Statistical Analysis 1: Comparison: MK-5442 5 mg vs Alendronate 70 mg; Test type: Superiority or Other; p < 0.001, Constrained Longitudinal Data Analysis — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = 187.31, 95% CI 2-sided [154.44 to 221.25]
Statistical Analysis 2: Comparison: MK-5442 7.5 mg vs Alendronate 70 mg; Test type: Superiority or Other; p < 0.001, Constrained Longitudinal Data Analysis — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = 200.29, 95% CI 2-sided [161.21 to 240.91]
Statistical Analysis 3: Comparison: MK-5442 10 mg vs Alendronate 70 mg; Test type: Superiority or Other; p < 0.001, Constrained Longitudinal Data Analysis — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = 224.30, 95% CI 2-sided [180.19 to 270.39]
Statistical Analysis 4: Comparison: Placebo vs MK-5442 5 mg; Test type: Superiority or Other; p = 0.034, Constrained Longitudinal Data Analysis — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = 48.29, 95% CI 2-sided [3.75 to 93.11]
Statistical Analysis 5: Comparison: Placebo vs MK-5442 7.5 mg; Test type: Superiority or Other; p = 0.019, Constrained Longitudinal Data Analysis — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = 61.27, 95% CI 2-sided [8.80 to 114.22]
Statistical Analysis 6: Comparison: Placebo vs MK-5442 10 mg; Test type: Superiority or Other; p = 0.002, Constrained Longitudinal Data Analysis — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = 85.28, 95% CI 2-sided [26.70 to 144.63]

13. Secondary Outcome: Least Squares Mean Percent Change From Baseline to Month 12 in Serum N-Terminal Propeptide (s-P1NP)
Description: s-P1NP is a sensitive marker of bone formation rate in the assessment of osteoporosis and is measured in units of ng/ml.
Time Frame: Baseline and Month 12
Population: as for outcome 11
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo | MK-5442 5 mg | MK-5442 7.5 mg | MK-5442 10 mg | Alendronate 70 mg
Number analyzed (Participants) | 70 | 73 | 69 | 73 | 71
percent change | 68.61 [51.82 to 87.27] | 127.18 [105.07 to 151.68] | 125.69 [102.92 to 151.01] | 163.96 [136.79 to 194.24] | -5.85 [-14.99 to 4.28]
Statistical Analysis 1: Comparison: MK-5442 5 mg vs Alendronate 70 mg; Test type: Superiority or Other; p < 0.001, Constrained Longitudinal Data Analysis — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = 133.03, 95% CI 2-sided [110.01 to 156.75]
Statistical Analysis 2: Comparison: MK-5442 5 mg vs Alendronate 70 mg; Test type: Superiority or Other; p = 0.001, Constrained Longitudinal Data Analysis — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = 133.03, 95% CI 2-sided [110.01 to 156.75]
Statistical Analysis 3: Comparison: MK-5442 7.5 mg vs Alendronate 70 mg; Test type: Superiority or Other; p < 0.001, Constrained Longitudinal Data Analysis — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = 131.53, 95% CI 2-sided [110.70 to 152.94]
Statistical Analysis 4: Comparison: MK-5442 10 mg vs Alendronate 70 mg; Test type: Superiority or Other; p < 0.001, Constrained Longitudinal Data Analysis — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = 169.80, 95% CI 2-sided [141.59 to 199.11]
Statistical Analysis 5: Comparison: Placebo vs MK-5442 5 mg; Test type: Superiority or Other; p < 0.001, Constrained Longitudinal Data Analysis — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = 58.57, 95% CI 2-sided [29.42 to 88.04]
Statistical Analysis 6: Comparison: Placebo vs MK-5442 7.5 mg; Test type: Superiority or Other; p < 0.001, Constrained Longitudinal Data Analysis — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = 57.07, 95% CI 2-sided [30.76 to 83.64]
Statistical Analysis 7: Comparison: Placebo vs MK-5442 10 mg; Test type: Superiority or Other; p < 0.001, Constrained Longitudinal Data Analysis — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = 95.34, 95% CI 2-sided [60.40 to 130.91]

14. Secondary Outcome: Least Squares Mean Percent Change From Baseline to Month 12 in Serum Bone-Specific Alkaline Phosphatase (s-BSAP)
Description: Bone Specific Alkaline Phosphatase is a biomarker of bone formation and is measured in units of μg/L.
Time Frame: Baseline and Month 12
Population: as for outcome 11
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo | MK-5442 5 mg | MK-5442 7.5 mg | MK-5442 10 mg | Alendronate 70 mg
Number analyzed (Participants) | 69 | 72 | 68 | 73 | 71
percent change | 29.51 [20.23 to 39.51] | 50.04 [39.60 to 61.25] | 49.98 [39.08 to 61.73] | 51.64 [40.42 to 63.76] | -3.83 [-10.41 to 3.24]
Statistical Analysis 1: Comparison: MK-5442 5 mg vs Alendronate 70 mg; Test type: Superiority or Other; p < 0.001, Constrained Longitudinal Data Analysis — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = 53.86, 95% CI 2-sided [39.31 to 68.60]
Statistical Analysis 2: Comparison: MK-5442 7.5 mg vs Alendronate 70 mg; Test type: Superiority or Other; p < 0.001, Constrained Longitudinal Data Analysis — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = 53.81, 95% CI 2-sided [41.37 to 66.38]
Statistical Analysis 3: Comparison: MK-5442 10 mg vs Alendronate 70 mg; Test type: Superiority or Other; p < 0.001, Constrained Longitudinal Data Analysis — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = 55.47, 95% CI 2-sided [41.19 to 69.94]
Statistical Analysis 4: Comparison: Placebo vs MK-5442 5 mg; Test type: Superiority or Other; p = 0.009, Constrained Longitudinal Data Analysis — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = 20.53, 95% CI 2-sided [5.96 to 35.03]
Statistical Analysis 5: Comparison: Placebo vs MK-5442 7.5 mg; Test type: Superiority or Other; p = 0.009, Constrained Longitudinal Data Analysis — [p-value comment as in outcome 1, analysis 1]; Difference in Least Mean Squares = 20.47, 95% CI 2-sided [5.96 to 35.03]
Statistical Analysis 6: Comparison: Placebo vs MK-5442 10 mg; Test type: Superiority or Other; p = 0.009, Constrained Longitudinal Data Analysis — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = 22.13, 95% CI 2-sided [4.47 to 39.89]

15. Secondary Outcome: Least Squares Mean Percent Change From Baseline to Month 12 in Serum Osteocalcin
Description: Serum osteocalcin is a biomarker of bone formation and is measured using units of nanograms (ng) / milliliter
  (mL).
Time Frame: Baseline and Month 12
Population: Analysis of osteocalcin was not conducted when it was determined that the efficacy of MK-5442 was not significantly different than placebo.
Arm/Group | Placebo | MK-5442 5 mg | MK-5442 7.5 mg | MK-5442 10 mg | Alendronate 70 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

16. Primary Outcome: Number of Participants With Trough Serum Calcium Level Exceeding Predefined Limits At Least Once
Description: Normal serum calcium level is 8-10 mg/dL (2-2.5 mmol/L) with some interlaboratory variation in the reference range, and hypercalcemia is defined as a serum calcium level greater than 10.5 mg/dL (>2.5 mmol/L).
  Based on these references, ≥10.6 mg/dL was predefined in this study as the cut-off for the normal limits of change. Participants with at least a one calcium level value ≥10.6 mg/dL were considered as having a "Tier 1" adverse event (AE). A Tier 1 AE was an AE of special interest identified a priori that could be used for inferential testing for statistical significance for between-group comparisons.
Time Frame: Baseline through Month 12
Population: All Participants as Treated (APaT): all randomized participants who received at least one dose of study treatment.
Measure: Number; unit: Participants
Groups:
- MK-5442 15 mg: Participants were initially randomized to receive oral, once-daily MK-5442 15 mg and once-weekly matching placebo to alendronate for 12 months.
  The MK-5442 15-mg treatment arm was discontinued as a result of Amendment 1 and thus no outcome analyses were performed.
Arm/Group | Placebo | MK-5442 5 mg | MK-5442 7.5 mg | MK-5442 10 mg | MK-5442 15 mg | Alendronate 70 mg
Number analyzed (Participants) | 88 | 87 | 88 | 87 | 88 | 84
Participants
  ≥10.6 ng/mL | 3 | 16 | 19 | 27 | 39 | 7
  ≥11.1 ng/mL | 1 | 1 | 4 | 7 | 19 | 1
  ≥12.1 ng/mL | 0 | 0 | 0 | 1 | 1 | 0

17. Primary Outcome: Number of Participants With Trough Albumin-Corrected Calcium Level Exceeding Predefined Limits At Least Once
Description: Albumin-Corrected Calcium = ([4 - plasma albumin in g/dL] × 0.8 + serum calcium).
  ≥10.6 mg/dL was predefined in this study as the cut-off for the normal limits of change. Participants with at least one albumin-corrected calcium level value ≥10.6 mg/dL were considered as having a "Tier 1" AE (an AE of special interest identified a priori that could be used for inferential testing for statistical significance for between-group comparisons).
Time Frame: Baseline through Month 12
Population: All Participants as Treated (APaT): all randomized participants who received at least one dose of study treatment.
Measure: Number; unit: Participants
Arm/Group | Placebo | MK-5442 5 mg | MK-5442 7.5 mg | MK-5442 10 mg | MK-5442 15 mg | Alendronate 70 mg
Number analyzed (Participants) | 88 | 87 | 88 | 87 | 88 | 84
Participants
  ≥10.6 ng/mL | 1 | 3 | 7 | 13 | 28 | 2
  ≥11.1 ng/mL | 1 | 0 | 1 | 3 | 9 | 0
  ≥12.1 ng/mL | 0 | 0 | 0 | 1 | 0 | 0

18. Primary Outcome: Number of Participants With Predefined Tier 1 Adverse Events
Description: Osteonecrosis of the jaw (ONJ), kidney stones, and bone neoplasms were predefined Tier-1 AEs in the study (an AE of special interest identified a priori that could be used for inferential testing for statistical significance for between-group comparisons).
Time Frame: Baseline through Month 12
Population: All Participants as Treated (APaT): all randomized participants who received at least one dose of study treatment.
Measure: Number; unit: Participants
Arm/Group | Placebo | MK-5442 5 mg | MK-5442 7.5 mg | MK-5442 10 mg | MK-5442 15 mg | Alendronate 70 mg
Number analyzed (Participants) | 88 | 87 | 88 | 87 | 88 | 84
Participants
  Osteonecrosis of the jaw | 0 | 0 | 0 | 0 | 0 | 0
  Kidney stones | 3 | 0 | 0 | 0 | 0 | 1
  Bone neoplasms | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Description: All Participants as Treated (APaT); all randomized participants who received at least one dose of study treatment.
Arm/Group | Placebo | MK-5442 5 mg | MK-5442 7.5 mg | MK-5442 10 mg | MK-5442 15 mg | Alendronate 70 mg
Serious Adverse Events (participants affected / at risk) | 6/88 | 5/87 | 4/88 | 6/87 | 4/88 | 1/88
Other Adverse Events (participants affected / at risk) | 18/88 | 18/87 | 26/88 | 32/87 | 28/88 | 10/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=88) | MK-5442 5 mg (N=87) | MK-5442 7.5 mg (N=88) | MK-5442 10 mg (N=87) | MK-5442 15 mg (N=88) | Alendronate 70 mg (N=88)
Angina Pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary Heart Disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertensive Heart Disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tako-Tsubo Cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis Eosinophilic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hernia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biliary Fistula (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Campylobacter Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Postoperative Pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postoperative Wound Complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Radius Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Foot Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Low Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cancer of the Head of the Pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Latigo Maligna Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carotid Artery Stenosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral Thrombosis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Migraine with Aura (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety Aggravated (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary Thromboembolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=88) | MK-5442 5 mg (N=87) | MK-5442 7.5 mg (N=88) | MK-5442 10 mg (N=87) | MK-5442 15 mg (N=88) | Alendronate 70 mg (N=84)
Constipation (Gastrointestinal disorders) | 3 (3) | 1 (1) | 5 (5) | 3 (4) | 1 (1) | 2 (2)
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 5 (5) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Urinary Tract Infection (Respiratory, thoracic and mediastinal disorders) | 5 (9) | 8 (10) | 6 (9) | 6 (8) | 2 (2) | 5 (6)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 8 (8) | 10 (12) | 23 (23) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 1 (1) | 8 (8) | 2 (2) | 1 (1)
Knee Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 6 (6) | 3 (3) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 7 (7) | 1 (1) | 2 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less